CLINICAL TRIAL: NCT03985137
Title: Role of the Balano-preputial Furrow 's Microbiota, in Circumcised Patients or Not, in the Acquisition or Transmission of HIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-24
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-infected patients: Male patient presenting at a follow-up consultation for HIV infection or following a Sexual Viral Exposure (EVA) accident, pre-exposure prophylaxis (PrEP) or screening for a Sexually Transmitted Infection (IST).
  Interventions: Other: mucocutaneous sampling by swab at the balano-preputial furrow.

INTERVENTIONS:
Other: mucocutaneous sampling by swab at the balano-preputial furrow. — the sample is made by the patient

SUMMARY:
The human immunodeficiency virus (HIV) remains at the moment a major public health problem. The figures currently report 37 million people infected with HIV worldwide, as well as 2 million new infections every year, the majority of which are men who have sex with men (MSM).

HIV research has accounted for more than 335,000 publications on PubMed since its first description in 1981. However, many questions remain unanswered, especially regarding the risk factors and protective factors, its transmission and acquisition, during sexual intercourse. By creating a background on PubMed with the keyword "HIV", we can see that at the end of the 80's, it was already established that male circumcision decreased the risk of transmission of HIV by 50 to 60%. Multiple hypotheses have been studied to justify this discovery, such as the reduction of micro-traumatisms, the modification of keratinization, the modification of penile anatomy induced by foreskin removal. In parallel, the rise of the study of the human microbiota, which refers to all microorganisms (bacteria, viruses, archaea, fungi and parasites) living in a specific environment, the human body, and this in a healthy or pathological situation. There is evidence that the microbiota may be involved in the pathogenesis of various diseases and may play a major role in the homeostasis of the human body. This implication has also interested researchers in the field of HIV : the protective role of circumcision in the acquisition and transmission of HIV has therefore begun to be studied in terms of the modification of the penile microbiome.

The first studies showed that circumcision had an impact on the abundance of bacteria present in the penis in humans, and modified the aerobic / anaerobic ratio in favor of the increase of aerobic bacteria. The first hypothesis was that circumcision played a protective role in the acquisition and transmission of HIV through a decrease in the diversity of the penile microbiota and in particular anaerobes.

This discovery was disrupted by the emergence of studies tending to question a microbiota predisposing to the risk of HIV acquisition in both men and women.

Indeed, it has been shown that certain bacteria (Prevotella, Dialister, ...) could favor the acquisition of the virus by the attraction in their wake of inflammation cells such as CD4 and Langerhans cells which would facilitate by their presence. , the penetration of the virus. This hypothesis has been proven in studies of bacterial vaginosis, which is known to be a risk factor for HIV acquisition and transmission. In 2012, results showed that the loss of Lactobacillus, in favor of anaerobic increases such as Gardnerella, Atopobium, and Prevotella, increased this risk against the HIV virus. Similarly, 7 bacteria have recently been incriminated in this phenomenon of susceptibility to HIV acquisition (Parvimonas, Gemella asaccharolytica, Mycoplasma hominis, Leptotrichia / Sneathia, Eggerthellaspecies and Megasphaeraspecies).Being committed to the exploration of the human microbiota in particular by culture, we propose to extend the knowledge of balano-preputial furrow 's microbiota in patients infected by HIV or not and supported in department Infectious Diseases. It is in this context, that a preliminary study carried out at the IHU between January and July 2018 made it possible to describe the existence of variability of the microbiota according to various criteria such as circumcision, HIV infection and sexual practices.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (18 years).
* Male patient presenting at a follow-up consultation for HIV infection or following a Sexual Viral Exposure (EVA) accident, pre-exposure prophylaxis (PrEP) or screening for a Sexually Transmitted Infection (IST).
* Person and / or legal guardian who has been informed of the study and has not expressed opposition to participate.
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* Person having expressed his opposition to participate in the study.
* Vulnerable person: person under tutorship or curatorship, or deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participation of a patient in the study requires only one visit. This visit will take place during a medical consultation at the "Infectious and Tropical Diseases" department for one of the following reasons:
  * HIV treatment follow-up;
  * Sexual AEV follow-up;
  * STI Screening
  * Follow-up of ARV treatment under PrEP.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
prevalence rate of bacteria | 12 months
  To compare the prevalence rate of bacteria between circumcised and uncircumcised patients by HIV or non-HIV status

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP HM
Locations (1):
- APHM, Marseille, Cedex 5, France